CLINICAL TRIAL: NCT03921749
Title: Radial Versus Focused Extracorporeal Shock Wave in the Treatment of Knee Osteoarthritis : A Randomized Control Trial
Brief Title: Radial Versus Focused Extracorporeal Shock Wave in the Treatment of Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Gwo-Chi Hu,PHD, Head of Physical Medicine and Rehbilitation, Associate Professor, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17MMHIS195
Record Dates: First submitted 2019-04-14; First posted 2019-04-19 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: group A : focused shock wave, group B: focused shock wave
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focused shock wave (Experimental): The extracorporeal shock wave will be applied to the patellofemoral and tibiofemoral borders and the subchondral bone of the medial tibia condyle of the affected knee joint. The intensities used will be focused shock wave therapy (0.20 mJ/mm 2 )
  Interventions: Device: Shockwave
- Raidal shock wave (Experimental): The extracorporeal shock wave will be applied to the patellofemoral and tibiofemoral borders and the subchondral bone of the medial tibia condyle of the affected knee joint. The intensities used will be radial shock wave therapy (3 bar)
  Interventions: Device: Shockwave

INTERVENTIONS:
Device: Shockwave — Both shockwave interventions will be administered without local anaesthesia. Three sessions will be administered at one-week intervals. During each session, 2000 pulses (1000 shots at the patellofemoral and tibiofemoral borders of the target knee and 1000 shots on the subchondral bone of the medial tibia condyle of the affected knee) will be delivered at 5 Hz. Energy flux density was 0.20 mJ/mm2 for patients in the "focused" group while "radial" shock waves were transmitted with 0.17 mJ/mm2 corresponding to a 3-bar energy level setting.

SUMMARY:
Radial versus Focused Extracorporeal Shock Wave in the Treatment of Knee Osteoarthritis : A Randomized Control Trial

DETAILED DESCRIPTION:
Background Knee Osteoarthritis (OA) is the most prevalent of the chronic rheumatic diseases and is a leading cause of pain and disability in most countries worldwide. The treatment methods for knee OA are diverse for patients with mild or moderate osteoarthritis (OA). Biomechanical intervention, physical therapy and exercise, medication, and intra-articular injections (both corticosteroid and hyaluronic acid) are recommended.

Recent studies have suggested that extracorporeal shock wave therapy is an effect treatment method for the knee OA. Based on the propagation pattern of the wave, extracorporeal shock wave therapy can be classified into two main modalities: focused and radial shock wave therapy. However, no previous study compared the effect of radial versus focused type of extracorporeal shock wave on symptoms and functions in patients with symptomatic knee OA. Therefore, the purpose of our study was to compare the effects of focused and radial shock wave therapy on patients with knee OA. Design: Randomized control trial Setting: Outpatient rehabilitation clinic in our hospital. Population:100 patients with mild and moderate knee OA Methods: Patients were randomly assigned to receive three sessions of either focused or radial shock wave therapy at 1-week intervals. The extracorporeal shock wave will be applied to the patellofemoral and tibiofemoral borders and the subchondral bone of the medial tibia condyle of the affected knee joint. The intensities that were used during focused shock wave therapy (0.20 mJ/mm 2 ) and radial shock wave therapy (3 bar) were comparable. The patients were evaluated at baseline and at 1, 4, and 8 weeks and 6 nmonths after the final shockwave treatment. The primary outcome measure was visual analogue scale. The secondary outcome measures were Western Ontario and McMaster Universities Osteoarthritis Index, the knee joint ROM, and sonographic findings and six-minute walk test (6MWT) will be performed. A linear mixed model with repeated measures was used to compare each outcome measure between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* people aged 45 years or more
* subjects diagnosed with knee OA according to the clinical criteria of the American College of Rheumatology
* subjects diagnosed with grade II or III OA during radiologicalexamination as defined by the radiological classification of Kellgren and Lawrence (K-L) scale for knee OA
* subjects with tenderness in the medial tibial plateau area
* subjects who had pain on one side of the knee.

Exclusion Criteria:

* patients with a history of spinal stenosis, evidence of neurologic disease by history or physical examination, or secondary causes of arthritis (inflammatory or metabolic)
* those who had a surgical intervention or intra-articular injection in the affected knee in the previous 6 months
* any contraindication to extracorporeal shock wave(pregnancy, cancer, coagulation disorders, inflammatory disease, pacemakers, or other electronic implants).

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-20 (Estimated); Primary Completion 2020-04-20 (Estimated); Study Completion 2020-05-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | The evaluation will be done before therapy sections, 1 week after, 4weeks and 8 weeks and 6 months after 3rd section of therapy.
  The scores will be based on pain intensity, where 0 and 10 points represent an absence of pain and a maximal intensity level of pain, respectively.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index | (6MWT). The evaluation will be done before therapy sections, 1 week after, 4weeks and 8 weeks and 6 months after 3rd section of therapy.
  The WOMAC, a validated disease-specific self-reporting questionnaire, is an examination for evaluating OA symptoms. The index consists of five questions for severity of knee pain, two for stiffness, and 17 for limitations in physical function. The WOMAC score ranges from 0 (best) to 96 (worst), with high score representing worse symptom severity31.
Lequesne index | The evaluation will be done before therapy sections, 1 week after, 4weeks and 8 weeks and 6 months after 3rd section of therapy.
  The Lequesne Index is a 10-question survey given to patients with osteoarthritis of the knee.
Six-minute walk test (6MWT) | The evaluation will be done before therapy sections, 1 week after and 8 weeks after 3rd section of therapy.
  Mobility performance will be assessed with the Six-Minute Walk Test (6MWT). The 6MWT is a submaximal test of walking capacity.33 Participants will walk at a self- selected speed for 6 min on an indoor, 30 meter corridor or walkway with cones placed at the beginning and end of the 30 meter boundary to indicate turns, with the goal of traveling the maximum distance. Jogging and running will not be allowed.
Measurement of knee ROM | The evaluation will be done before therapy sections, 1 week after and 8 weeks after 3rd section of therapy.
  The assisted active ROM will be measured using a hand-held goniometry.Measurements of knee flexion and extension will be taken with patients lying supine on an examination couch. The fully extended knee is considered as the zero position, and the degrees of maximum flexion, maximum extension, and extension deficit, when present, will be recorded. A negative ROM score for extension indicated that the patient is unable to reach the zero position. The angle between maximum flexion and maximum extension will be described as the excursion range.

CONTACTS AND LOCATIONS:
Overall Officials: Gwo Chi Hu, Principal Investigator — Taiwan Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ko NY, Chang CN, Cheng CH, Yu HK, Hu GC. Comparative Effectiveness of Focused Extracorporeal versus Radial Extracorporeal Shockwave Therapy for Knee Osteoarthritis-Randomized Controlled Study. Int J Environ Res Public Health. 2022 Jul 24;19(15):9001. doi: 10.3390/ijerph19159001. PMID 35897371